CLINICAL TRIAL: NCT05017077
Title: Home Telemonitoring in Pediatric Heart Failure
Brief Title: Home Monitoring in Pediatric Heart Failure
Acronym: HOPE-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Rachele Adorisio, Principal Investigator, Bambino Gesù Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2240_OPBG_2020
Record Dates: First submitted 2021-03-11; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Pediatric Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemonitoring (Experimental): To evaluate the feasibility and efficacy of a new model of tele monitoring in pediatric population in advanced heart failure, we will enroll 20 patients in advanced NYHA/Ross class in waiting list for Heart Transplant. An home telemonitoring capable to detect vital parameters as heart rate, body temperature, blood pressure, oxygen saturation, breathe frequency, weight, arrhythmias and cardiac index may offers to physician valuable information able to strictly monitoring the clinical status of patients
  Interventions: Device: DynaVision System

INTERVENTIONS:
Device: DynaVision System — Telemonitoring for pediatric heart failure

SUMMARY:
Heart failure is a complex clinical syndrome, representing the final evolution of many cardiac diseases that may differ for etiology and pathophysiology. In pediatric population, it is particularly challenging to manage because of the heterogeneity in age, primary cardiac disease, and the broad range of clinical signs and symptoms. Frequent hospitalizations are current problem. Hospitalization within the first year since the first episode, lack of adherence to medical therapy and diet difficulties are the main issues in this population of patients, and they rebounds on prognosis and public health costs. Actions aimed to prevent and manage these matters will improve outcome in patients with chronic heart failure. Telemedicine proved its usefulness in adult population, but, nowadays, no studies have been conducted in children. From the beginning of 21th century, remote monitoring attempts have been adopted, initially by phone calls. Currently, the e-care monitoring fits in the context of telemedicine 2.0 based on new communication models. The aim of this study is to affirm the feasibility and efficacy of a new model of tele monitoring in pediatric population. High-risk patients need a strict clinical control normally difficult to adopt. A telematics system capable to detect vital parameters as heart rate, body temperature, blood pressure, oxygen saturation, breathe frequency, weight, arrhythmias and cardiac index may offers to physician valuable information able to strictly monitoring the clinical status of patients. All of these data permits to physician to early detect critical signals of a deteriorated status, modify adherence to care and implement therapeutic strategies in order to prevent frequent hospitalizations. Our project provides a system of continuous tele-monitoring of vital parameters through a patch applied on the chest of the baby. Data are sent to a service center, "virtual clinic" and daily analyzed in multiparametric system by a specialized nurse. On the basis of pre-established alarms, the virtual clinic will notify to physician. Feasibility and tolerability of this new monitoring system will be evaluated after a 3 months period on a cohort of 20 patients affected by chronic, high-risk, heart failure.

ELIGIBILITY:
Inclusion Criteria:

* NYHA/Ross class III or IV
* Severe impairment of ventricular function (EF < 40%) both for left or univentricular
* Prior hospitalization for acute heart failure within 1 year
* At least 2 prior hospitalization for acute heart failure
* Patients on waiting list for orthotopic heart transplantation (UNOS 1B,2)
* Informed consent obtained

Exclusion Criteria:

* PMK or ICD
* hospitalized patients
* neurological or psychiatric impairment
* urgent waiting list for heart transplantation (UNOS 1A)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | three months
  number of day (percentage) of adherence to telemonitoring, at least 18 hours per day when the patient kept the patch applied at 3 months.

SECONDARY OUTCOMES:
Number of hours of patch kept applied | at 1 week
  Tolerability
Number of hours of patch kept applied | at 3 months
  Tolerability
Interquartile Range - median of hours of patch kept applied | at 1 week
  Tolerability
Interquartile Range - median of hours of patch kept applied | at 3 months
  Tolerability
Number of unplanned hospitalization | 3 months
  Reliability
Number of life treating arrhythmias | 3 months
  Reliability
Mortality | 3 months
  Reliability
Number of unplanned hospital access (day hospital / ambulatory) | 3 months
  Reliability
Comparison to levels of Hemoglobin (g/dL) | 3 months
  Reliability
Comparison to levels of Albumin (g/dL) | 3 months
  Reliability
Comparison to levels of Sodium (mEq/L) | 3 months
  Reliability
Comparison to levels of Potassium (mEq/L) | 3 months
  Reliability
Comparison to levels of Serum Creatinine (mg/dL) | 3 months
  Reliability
Satisfaction questionnaire | 1 week
  Satisfaction
Satisfaction questionnaire | 3 months
  Satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Bambino Gesù Hospital, Rome, Italy